CLINICAL TRIAL: NCT00341510
Title: U.S. Health Behavior in School Children Survey
Brief Title: Health Behaviors in School-age Children: A World Health Organization Cross-National Study
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906017; 06-CH-N017
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-11-28

CONDITIONS: Health Behavior
Keywords: Risk Behavior; Health Status; Adolescence; Positive Health Behaviors; Social Support; Health Behavior; Survey
MeSH Terms: conditions — Health Behavior; Risk-Taking

SUMMARY:
This study is a survey (Health Behaviors in School-age Children) sponsored by the World Health Organization to gather information about nutrition, dieting practices, physical activity, injuries, violence, relationships with family and friends, perceptions of school as a supportive environment, alcohol and tobacco use and drug use among adolescents, and about the communities in which students live. The U.S. sponsors of the survey are the National Institutes of Health and the Health Resources and Services Administration.

The objectives of the international HBSC study are:

* To assess the prevalence of early adolescent health behaviors
* To identify psychosocial factors associated with adolescent behaviors
* To provide an opportunity for analyses of cross-national comparisons
* To provide an opportunity for analyses of trends in the U.S. and cross-nationally

In addition to the above, the survey includes additional questions designed to provide information about areas of specific national interest, including the following:

* To assess the association of school, family, peers, and other environmental factors on health behavior and health status
* To assess the prevalence and identify factors associated with diet and physical activity
* To assess the prevalence and identify factors associated with bullying and risk behaviors.

This is the third U.S. administration of the HBSC survey, previously administered in 1997-1998 and 2001-2002.

U.S. participants in the survey include about 15,000 students from 350 schools selected to take part across the country. In each school, one or two classes (about 25 students) in each grade 6 through 10 are picked randomly to participate. In one class period, the students complete the written survey, which has 80 multiple choice questions. Students do not put their name on the survey. When they finish the survey, the place it in an envelope and seal it shut. The envelopes are then put in a box. Reports will not include the names of participating counties, cities, school districts, schools, or students.

The information collected from U.S. school children is compared with similar information collected from school children in 36 other countries. The survey is used to help set national priorities for school and youth programs, as well as to monitor the progress of these programs.

DETAILED DESCRIPTION:
The Health Behaviors in School-age Children (HBSC) survey is the only international survey of its type and the only national survey of adolescent health behavior in the U.S. The U.S. HBSC complements the Youth Risk Behavior Survey (YRBS) and the Monitoring the Future surveys of older adolescents. The aims of the survey are to assess the prevalence of health behaviors and identify factors associated with them in a national probability sample of 6th -10th grade students, allowing for trend analyses and cross-national comparisons among the 37 countries involved in the quadrennial international HBSC surveys. This would be the third U.S. administration of the HBSC survey, previously administered in 1997-1998 and 2001-2002.

ELIGIBILITY:
-INCLUSION CRITERIA:

6th and 10th grade students

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14350
Dates: Start 2005-10-17; Study Completion 2006-11-28

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

REFERENCES:
- [Background] Simons-Morton BG, Hartos JL, Haynie DL. Prospective analysis of peer and parent influences on minor aggression among early adolescents. Health Educ Behav. 2004 Feb;31(1):22-33. doi: 10.1177/1090198103258850. PMID 14768655